CLINICAL TRIAL: NCT05669105
Title: Prospective Collection of Whole Blood From Active Non-Small Cell Lung Cancer Patients for Supplemental Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-08877
Record Dates: First submitted 2022-12-13; First posted 2022-12-30 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Specimen sample — Participants will have up to 100 mL of whole blood collected.

SUMMARY:
The study objective is to collect biospecimen samples (e.g., whole blood) from participants diagnosed with active lung cancer to investigate the immune response to develop treatments and therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to provide written informed consent
* Participants are willing and able to provide appropriate photo identification
* Participant's age 18 - 100 years old
* Participants diagnosed with active non-small cell lung cancer (Adenocarcinoma or Squamous Cell only. All stages are acceptable.)
* Participants must have associated tissue biomarker data (EFGR and MET mutations) in their medical records

Exclusion Criteria:

* Participants who are pregnant or nursing
* Participants with a known history of HIV, hepatitis, or other infectious diseases
* Participants who have taken an investigational product in the last 30 days
* Participants who have experienced excess blood loss, including blood donation defined as 250 mL in the last month or 500 mL in the previous two months
* Participants currently enrolled in a clinical trial
* Participants currently in remission

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 200 participants. Recruitment will occur through Sanguine advertisements, partnerships with cancer foundations, and cancer centers. Participants may be contacted for future studies.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-19 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Biospecimen & Clinical Data Collection | 10 years
  The primary objective is to collect 2000 whole blood samples from subjects who are diagnosed with active lung cancer.
  The purpose of this study is to collect biospecimen samples (e.g., whole blood) from participants diagnosed with various active lung cancers so that investigations can analyze how the immune response can take place, and aid in understanding active lung cancer biomarkers for future early diagnosis and treatment options.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine Biosciences, Waltham, Massachusetts, United States